CLINICAL TRIAL: NCT01286285
Title: An Active, Epidemiological Surveillance Study on Influenza-related Hospitalizations to Intensive Care Units and Fatalities in Paediatric Hospitals in Bavaria Covering the Influenza Seasons 2010/2011 and 2011/2012
Brief Title: Surveillance of Influenza in Paediatric Intensive Care Units in Bavaria
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Children's Hospital, Wuerzburg (Other)
Collaborators: GlaxoSmithKline (Industry); University of Wuerzburg (Other)
Responsible Party: Prof. Dr. med. Johannes G. Liese, MSc, University Children's Hospital Wuerzburg, Germany
Other Study IDs: UNIV HOSP WUERZBURG 7106877
Record Dates: First submitted 2011-01-19; First posted 2011-01-31 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Influenza; Acute Respiratory Infection
Keywords: influenza; acute respiratory infections; paediatric; intensive care units; epidemiology
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Naso-pharyngeal swab, if not available nasal wash or other respiratory secretion (only if collected routinely by the hospital)
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to assess the number of severe, laboratory-confirmed influenza in children hospitalized to paediatric intensive care units. Furthermore, the proportion of these children from all children hospitalized to paediatric intensive care units with acute respiratory infections will be established.

DETAILED DESCRIPTION:
Accurate epidemiological data on severe influenza-associated hospitalizations and fatalities in children are lacking in Germany. The purpose of this study is primarily, to assess the number of severe, laboratory-confirmed influenza in children hospitalized to paediatric intensive care units due to suspected acute respiratory infections/ influenza/ influenza-triggered complications and in children developing influenza during paediatric intensive care unit hospitalization, as well as the number of influenza-associated fatalities. In addition we aim at assessing clinical features, severity, risk factors, complications, diagnostic procedures, treatment and outcome of severe, laboratory-confirmed influenza (and other acute respiratory infections) in these children. Another objective is to estimate the proportion of laboratory-confirmed influenza cases in all children hospitalized to paediatric intensive care units with acute respiratory infections and to evaluate the number and proportion of paediatric intensive care unit hospitalizations due to other viral acute respiratory infections. Additional aims are to estimate the (minimum) incidence of severe influenza-associated hospitalizations in Bavarian children and to estimate the (minimum) incidences of other acute respiratory infections.

Ideally, this study will be conducted between October 2010 and March 2012 in all Bavarian (Germany) hospitals with paediatric intensive care units or paediatric intensive care beds (neonatology excluded). To optimize reporting there will be one study physician at each site responsible for documentation, diagnostic procedures and queries. The local study physician will receive an initiation visit at the start of each season, and will be contacted by the study coordination (situated at the University Children's Hospital in Wuerzburg) bi-weekly by phone. This local study physician summarizes the paediatric intensive care unit admittance in a log sheet, documents epidemiological, demographical, and clinical data in a questionnaire for all suspected acute respiratory infections/influenza patients with parental informed consent (pseudonymous data only), and draws a nasopharyngeal swab or -wash if indicated as routine procedure. A sample will be sent to the central laboratory (Institute for Virology and Immunobiology, University of Wuerzburg) for analysis (influenza-polymerase chain reaction, influenza virus subtyping, other viral acute respiratory infections (respiratory syncytial virus, parainfluenza 1-4, humane metapneumovirus, adenoviruses, rhinoviruses, enteroviruses). The central laboratory will analyse the samples timely and report the results to the respective study site. Additional influenza-tests may also be performed by the local laboratory, at the discretion of the hospitals. All tests, locally and performed in Wuerzburg, and their outcome should be reported in the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, ≤16 years of age at the time of paediatric intensive care unit admittance. A subject will become ineligible on his/her 17th birthday
* All patients for whom a written Informed Consent Form for study participation can be obtained
* Children presenting with suspected acute respiratory infection of the upper or lower respiratory tract, with acute respiratory infection-related symptoms, e.g. sore throat (in children ≥ 3 years old), coryza (runny nose), cough etc. or B) Children already admitted to the paediatric intensive care unit without apparent acute respiratory infection/influenza-related symptoms that develop acute respiratory infection/influenza-related symptoms within the paediatric intensive care unit or
* Children admitted to the paediatric intensive care unit with suspected influenza (even without respiratory symptoms, e.g. with neurological symptoms) or
* Children admitted to the paediatric intensive care unit with potential influenza-triggered complications and laboratory-confirmed influenza ≤14 days before paediatric intensive care unit admission (by polymerase chain reaction or other influenza test methods)
* Additionally, all children with confirmed / suspected acute respiratory infection/ influenza that died already during admission to the paediatric hospital/ the paediatric intensive care unit will be included (a pseudonymous autopsy report including laboratory analyses (if available) will be requested for these patients).

Exclusion Criteria:

none

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children ≤16 years of age, in hospitals with paediatric intensive care units or paediatric intensive care beds in Bavaria, Germany
Sampling Method: Non-Probability Sample
Enrollment: 1140 (Estimated)
Dates: Start 2010-10; Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
number and proportion of influenza-/ acute respiratory infection-associated hospitalizations to paediatric intensive care units | outcome measure will be assessed between March and June 2012 for the whole study period (October 2010 - March 2012)
  * To evaluate the number of laboratory-confirmed influenza-associated (seasonal and new influenza A (H1N1)) hospitalizations to paediatric intensive care units in children ≤16 years of age
  * To evaluate the proportion of laboratory-confirmed influenza-associated (seasonal and new influenza A (H1N1)) hospitalizations to paediatric intensive care units in all children ≤16 years of age hospitalized to paediatric intensive care units with acute respiratory infections or suspected influenza

SECONDARY OUTCOMES:
health status at discharge | outcome measure will be assessed between March and June 2012 for the whole study period (October 2010 - March 2012)
  - To evaluate the health status at discharge (outcome: alive without sequelae, alive with sequelae, deceased) in children ≤16 years of age hospitalized to paediatric intensive care units with laboratory-confirmed influenza (seasonal and new influenza A (H1N1))
severity of disease | outcome measure will be assessed between March and June 2012 for the whole study period (October 2010 - March 2012)
  - To evaluate the severity of disease in children ≤16 years of age hospitalized to paediatric intensive care units with laboratory-confirmed influenza (seasonal and new influenza A (H1N1))
symptoms and complications | outcome measure will be assessed between March and June 2012 for the whole study period (October 2010 - March 2012)
  * To evaluate the number of laboratory-confirmed influenza-associated (seasonal and new influenza A (H1N1)) cases treated with mechanical ventilation in children ≤16 years of age hospitalized to paediatric intensive care units
  * To evaluate symptoms, complications, risk factors, and therapeutic procedures in children ≤16 years of age hospitalized to paediatric intensive care units with laboratory-confirmed influenza (seasonal and new influenza A (H1N1))
comparison between influenza A and B as well as seasonal and new influenza | outcome measure will be assessed between March and June 2012 for the whole study period (October 2010 - March 2012)
  * To compare age distribution, symptoms, complications, severity, risk factors, therapeutic procedures and outcome (fatalities, sequelae) between seasonal influenza A (and subtypes) and influenza B (and lineages) in children ≤16 years of age hospitalized to paediatric intensive care units
  * To compare age distribution, symptoms, complications, severity, risk factors, therapeutic procedures and outcome (fatalities, sequelae) between seasonal influenza and new influenza A (H1N1) in children ≤16 years of age hospitalized to paediatric intensive care units
comparison of different influenza tests | outcome measure will be assessed between March and June 2012 for the whole study period (October 2010 - March 2012)
  - To evaluate the positive rate of other microbiological influenza tests than polymerase chain reaction (rapid test, immunoflourescence etc, if locally performed by hospitals/laboratories) in children ≤16 years of age hospitalized to paediatric intensive care units
number of acute respiratory infection-associated hospitalizations to paediatric intensive care units, comparison with influenza-associated hospitalizations to paediatric intensive care units | outcome measure will be assessed between March and June 2012 for the whole study period (October 2010 - March 2012)
  * To evaluate the number and proportion of hospitalizations to paediatric intensive care units admitted due to other acute respiratory infections in children ≤16 years of age
  * To compare age distribution, symptoms, complications, severity, risk factors, therapeutic procedures, and outcome (fatalities/sequelae) between children hospitalized to paediatric intensive care units with influenza and children hospitalized to paediatric intensive care units due to other acute respiratory infections
number of hospitalizations related to the corresponding population | outcome measure will be assessed between March and June 2012 for the whole study period (October 2010 - March 2012)
  * To estimate the (minimum) incidence of laboratory-confirmed influenza (seasonal and new influenza A (H1N1)) hospitalizations to paediatric intensive care units in Bavaria in children ≤16 years of age
  * To estimate the (minimum) incidence of laboratory-confirmed hospitalizations to paediatric intensive care units in Bavaria in children ≤16 years of age due to other acute respiratory infections

CONTACTS AND LOCATIONS:
Overall Officials: Johannes G. Liese, MD, MSc, Principal Investigator — University Children's Hospital Wuerzburg, Paediatric Infectiology and Immunology, Josef-Schneider-Str. 2, 97080 Wuerzburg, Germany
Locations (1):
- University Children's Hospital Wuerzburg, Würzburg, Bavaria, Germany

REFERENCES:
- [Background] Milne BG, Williams S, May ML, Kesson AM, Gillis J, Burgess MA. Influenza A associated morbidity and mortality in a Paediatric Intensive Care Unit. Commun Dis Intell Q Rep. 2004;28(4):504-9. doi: 10.33321/cdi.2004.28.58. PMID 15745400
- [Background] Poehling KA, Edwards KM, Weinberg GA, Szilagyi P, Staat MA, Iwane MK, Bridges CB, Grijalva CG, Zhu Y, Bernstein DI, Herrera G, Erdman D, Hall CB, Seither R, Griffin MR; New Vaccine Surveillance Network. The underrecognized burden of influenza in young children. N Engl J Med. 2006 Jul 6;355(1):31-40. doi: 10.1056/NEJMoa054869. PMID 16822994
- [Background] Rojo JC, Ruiz-Contreras J, Fernandez MB, Marin MA, Folgueira L. Influenza-related hospitalizations in children younger than three years of age. Pediatr Infect Dis J. 2006 Jul;25(7):596-601. doi: 10.1097/01.inf.0000220208.59965.95. PMID 16804428
- [Background] Finelli L, Fiore A, Dhara R, Brammer L, Shay DK, Kamimoto L, Fry A, Hageman J, Gorwitz R, Bresee J, Uyeki T. Influenza-associated pediatric mortality in the United States: increase of Staphylococcus aureus coinfection. Pediatrics. 2008 Oct;122(4):805-11. doi: 10.1542/peds.2008-1336. PMID 18829805
- [Background] Libster R, Bugna J, Coviello S, Hijano DR, Dunaiewsky M, Reynoso N, Cavalieri ML, Guglielmo MC, Areso MS, Gilligan T, Santucho F, Cabral G, Gregorio GL, Moreno R, Lutz MI, Panigasi AL, Saligari L, Caballero MT, Egues Almeida RM, Gutierrez Meyer ME, Neder MD, Davenport MC, Del Valle MP, Santidrian VS, Mosca G, Garcia Dominguez M, Alvarez L, Landa P, Pota A, Bolonati N, Dalamon R, Sanchez Mercol VI, Espinoza M, Peuchot JC, Karolinski A, Bruno M, Borsa A, Ferrero F, Bonina A, Ramonet M, Albano LC, Luedicke N, Alterman E, Savy V, Baumeister E, Chappell JD, Edwards KM, Melendi GA, Polack FP. Pediatric hospitalizations associated with 2009 pandemic influenza A (H1N1) in Argentina. N Engl J Med. 2010 Jan 7;362(1):45-55. doi: 10.1056/NEJMoa0907673. Epub 2009 Dec 23. PMID 20032320
- [Background] Kumar A, Zarychanski R, Pinto R, Cook DJ, Marshall J, Lacroix J, Stelfox T, Bagshaw S, Choong K, Lamontagne F, Turgeon AF, Lapinsky S, Ahern SP, Smith O, Siddiqui F, Jouvet P, Khwaja K, McIntyre L, Menon K, Hutchison J, Hornstein D, Joffe A, Lauzier F, Singh J, Karachi T, Wiebe K, Olafson K, Ramsey C, Sharma S, Dodek P, Meade M, Hall R, Fowler RA; Canadian Critical Care Trials Group H1N1 Collaborative. Critically ill patients with 2009 influenza A(H1N1) infection in Canada. JAMA. 2009 Nov 4;302(17):1872-9. doi: 10.1001/jama.2009.1496. Epub 2009 Oct 12. PMID 19822627
- [Background] Weigl JA, Puppe W, Schmitt HJ. The incidence of influenza-associated hospitalizations in children in Germany. Epidemiol Infect. 2002 Dec;129(3):525-33. doi: 10.1017/s0950268802007707. PMID 12558335